CLINICAL TRIAL: NCT03303092
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial Evaluating the Efficacy and Safety of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Episodic Migraine
Brief Title: Efficacy and Safety of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Episodic Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 406-102-00002; JapicCTI-173725 (Other: Japic)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEV-48125 (225/225/225 mg) group (Experimental): TEV-48125 will be subcutaneously administered once monthly for 3 months (225/225/225 mg).
  Interventions: Drug: TEV-48125
- TEV-48125 (675 mg/placebo/placebo) group (Experimental): TEV-48125 or placebo will be subcutaneously administered once monthly for 3 months (675 mg/placebo/placebo).
  Interventions: Drug: TEV-48125 or placebo
- Placebo group (Placebo Comparator): Placebo will be subcutaneously administered once monthly for 3 months (placebo/placebo/placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-48125 — TEV-48125 will be subcutaneously administered once monthly for 3 months.
  Arms: TEV-48125 (225/225/225 mg) group
Drug: TEV-48125 or placebo — TEV-48125 or placebo will be subcutaneously administered once monthly for 3 months.
  Arms: TEV-48125 (675 mg/placebo/placebo) group
Drug: Placebo — Placebo will be subcutaneously administered once monthly for 3 months.
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy and safety of subcutaneous (SC) administration of TEV-48125 (monthly TEV-48125 225 mg and TEV-48125 675 mg once over a period of 3 months) compared with placebo for preventive treatment in Episodic Migraine patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine (according to The International Classification of Headache Disorders, third edition [beta version] criteria) or clinical judgment suggests a migraine diagnosis
* Patient fulfills the criteria for Episodic migraine in baseline information collected during the 28 day screening period
* Not using preventive migraine medications for migraine or other medical conditions or using no more than 1 preventive migraine medication for migraine or other medical conditions if the dose and regimen have been stable for at least 2 months prior to giving informed consent.
* Patient demonstrates compliance with the electronic headache diary during the screening period by entry of headache data on a minimum of 24 of 28 days and the entered data is judged appropriate by the investigator.

Exclusion Criteria:

Patients who have previously failed (lack of efficacy) 2 or more of the clusters of the medications for treatment of migraine after use for at least 3 months at accepted migraine therapeutic doses

- Hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, or ocular disease considered clinically significant in the judgment of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Saitama Medical University Hospital, Iruma, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Takeshima T, Nakai M, Shibasaki Y, Ishida M, Kim BK, Ning X, Koga N. Early onset of efficacy with fremanezumab in patients with episodic and chronic migraine: subanalysis of two phase 2b/3 trials in Japanese and Korean patients. J Headache Pain. 2022 Feb 9;23(1):24. doi: 10.1186/s10194-022-01393-0. PMID 35139816

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Started | 121 | 119 | 117
Completed | 118 | 113 | 112
Not Completed | 3 | 6 | 5
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 5 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group | Total
Number analyzed (Participants) | 121 | 119 | 117 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 116 | 112 | 348
  >=65 years | 1 | 3 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (9.5) | 41.9 (10.1) | 44.2 (10.7) | 43.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 101 | 100 | 302
  Male | 20 | 18 | 17 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 121 | 119 | 117 | 357
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 102 | 101 | 98 | 301
  South Korea | 19 | 18 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Monthly (28 Days) Average Number of Migraine Days During the 12-week Period After the First Dose of Investigational Medicinal Product (IMP)
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, the subjects were asked to enter headache data in the electronic headache diary for the previous 24-hour period.
  Subjects who reported headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications).
  Overall headache duration was recorded numerically, in hours, as well as number of hours with headache of at least moderate severity.
  If headache was reported, then headache severity was subjectively rated by the subject as follows: Mild headache, Moderate headache, Severe headache. Subjects also recorded the presence or absence of photophobia, phonophobia, nausea, or vomiting, and the status of use of any acute headache medications.
Time Frame: Baseline, 12 weeks
Population: Full Analysis set (FAS): Subjects who received the IMP at least once and had baseline and Week 12 data on monthly average number of migraine days.
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 121 | 117 | 116
days/month | -4.00 (0.37) | -4.02 (0.38) | -1.02 (0.38)

2. Secondary Outcome: Proportion of Subjects Reaching at Least 50% Reduction in the Monthly Average Number of Migraine Days During the 12-week Period After the First Dose of IMP
Description: as for outcome 1
Time Frame: 12 weeks
Population: Full Analysis set (FAS): Subjects who received the IMP at least once and had baseline and Week 12 data on monthly average number of migraine days. "Overall Number of Participants Analyzed" = the number of subjects meeting responder criteria.
Measure: Number; unit: percentage of participants
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 50 | 53 | 13
percentage of participants | 41.3 | 45.3 | 11.2

3. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of Days With Use of Any Acute Headache Medications During the 12-week Period After the First Dose of IMP
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, subjects entered headache data in the electronic headache diary for the previous 24-hour period. Subjects who reported headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications).
Time Frame: Baseline, 12 weeks
Population: Full Analysis set (FAS): Subjects who received the IMP at least once and had baseline and Week 12 data on monthly average number of migraine days. "Overall Number of Participants Analyzed" = the number of subjects with both baseline and assessment at each visit.
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 121 | 117 | 116
days/month | -3.30 (0.34) | -3.29 (0.36) | -0.46 (0.35)

4. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of Migraine Days During the 12-week Period After the First Dose of IMP in Patients Not Receiving Concomitant Preventive Migraine Medications
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 97 | 94 | 94
days/month | -4.42 (0.36) | -4.21 (0.37) | -1.40 (0.37)

5. Secondary Outcome: Mean Change From Baseline in Disability Score, as Measured by Migraine Disability Assessment (MIDAS) Questionnaire at 4 Weeks After the Final (Third) Dose of IMP
Description: Using the MIDAS questionnaire, subjects assessed the degree of headache-related disability based on lost days of activity in 3 domains (work, household work, and nonwork) over the last 3 months. The MIDAS questionnaire was a 5-item instrument. The total of the scores of the first 5 questions was used for grading the level of disability, with scores of 0 to 5, 6 to 10, 11 to 20, and ≥ 21 interpreted as disability grades I (little or no disability), II (mild disability), III (moderate disability), and IV (severe disability), respectively.
Time Frame: Baseline, 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 118 | 112 | 112
score on a scale | -12.64 (1.42) | -12.55 (1.49) | -7.41 (1.46)

ADVERSE EVENTS:
Time Frame: Double-blind treatment period (12 weeks)
Description: Safety set (SS):Subjects who received the IMP at least once.
Arm/Group | TEV-48125 (225/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/118 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/118 | 0/117
Other Adverse Events (participants affected / at risk) | 69/121 | 74/118 | 77/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEV-48125 (225/225/225 mg) Group (N=121) | TEV-48125 (675 mg/Placebo/Placebo) Group (N=118) | Placebo Group (N=117)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Purpura non-thrombocytopenic (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 19 | 14 | 15
Injection site induration (General disorders) | 18 | 14 | 12
Injection site pain (General disorders) | 11 | 16 | 7
Injection site pruritus (General disorders) | 7 | 2 | 0
Injection site swelling (General disorders) | 4 | 2 | 0
Injection site rash (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0
Injection site dermatitis (General disorders) | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 4 | 1
Injection site macule (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site eczema (General disorders) | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1
Injection site urticaria (General disorders) | 0 | 1 | 0
Injection site warmth (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 17 | 15 | 16
Influenza (Infections and infestations) | 6 | 2 | 1
Bacterial vulvovaginitis (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Occult blood positive (Investigations) | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 4
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Vascular headache (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 3
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tumour excision (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03303092/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT03303092/SAP_001.pdf